CLINICAL TRIAL: NCT06782542
Title: Single-Arm Phase 2 Study of Olutasidenib, Venetoclax, and Azacitidine in IDH1 Mutated Newly Diagnosed Acute Myeloid Leukemia Patients Who Are Eligible for Intensive Induction Chemotherapy
Brief Title: Olutasidenib, Venetoclax, and Azacitidine in IDH1 Mutated Newly Diagnosed Acute Myeloid Leukemia Patients Eligible for Intensive Induction Chemotherapy
Acronym: OLUVENAZA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Justin Watts, MD (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Justin Watts, MD, Associate Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240763
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; IDH1 Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — olutasidenib; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OLUVENAZA Treatment Group (Experimental): Participants in this group will receive combination treatment of Olutasidenib, Venetoclax and Azacitidine orally for up to 12 cycles, each cycle lasting 28 days. Total participation duration is about 14 months
  Interventions: Drug: Olutasidenib; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Olutasidenib — Olutasidenib will be supplied as 150 mg capsules to be administered orally, twice per day (BID) on an empty stomach (fasting at least 1 hour before or 2 hours after a meal), starting on Cycle 1 Day 1, and will be given continuously.
Drug: Venetoclax — Participants will receive Venetoclax as a 100mg tablet to be self-administered orally with a meal and water once daily, two hours after starting Olutasidenib administration, starting on Cycle 1 Day 1. The dosing regimen of Venetoclax is as follows:
  * Cycle 1: Days 1 - 21 over a 28-day cycle
  * Cycle 1 Week 1: Ramp-up dosing schedule up to 400mg (4 x 100mg/tablet)
  * For participants with blast clearance: Cycle 2 and beyond: Days 1 - 14 over a 28-day cycle
  * For participants with persistent clearance: Cycle 2 through 4: Days 1 - 21
Drug: Azacitidine — Participants will receive Azacitidine 75 mg/m2 per day via subcutaneous (SC) injection or intravenous (IV) infusion on Days 1-7 of each cycle.

SUMMARY:
The purpose of this study is as follows:

1. Determine whether people receiving the combination treatment of olutasidenib, venetoclax, and azacitidine have the same, more, or fewer side effects compared to the usual chemotherapy treatment that people with this condition receive.
2. Determine how well the combination treatment of olutasidenib, venetoclax, and azacitidine works compared to the usual chemotherapy treatment that people with this condition receive.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is an adult male or female participant aged 18-75 years considered eligible to undergo intensive induction chemotherapy at the time of signing the informed consent form (ICF).
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
3. Confirmed diagnosis of:

   1. Newly diagnosed AML Isocitrate dehydrogenase 1 (IDH1) R132 mutated disease as assessed locally. Note: historical results from within 30 days of informed consent will be accepted if the participant did not receive systemic treatment after collection.
   2. Secondary AML, including prior hypomethylating agents (HMA) exposure for myelodysplastic syndrome (MDS), myeloproliferative neoplasms (MPN), or MDS/MPN is allowed.
4. Participant must have adequate organ function, defined by the following:

   1. Aspartate transaminase (AST) and alanine aminotransferase (ALT) values ≤3 × upper limit of normal (ULN) or ≤5 × ULN for participants with leukemic involvement.
   2. Bilirubin ≤2 ULN (≤3 × ULN in participants with Gilbert Syndrome) or ≤3 × ULN for participants with leukemic involvement.
   3. Creatinine clearance ≥30 mL/min (using Cockcroft-Gault), or serum creatinine ≤1.5 × ULN.
5. The interval from prior treatment for an antecedent hematologic disorder to the first dose of study treatment (C1D1) will be at least 7 days for cytotoxic or non-cytotoxic (immunotherapy) agents. In addition, the following will be allowed:

   1. Intrathecal chemotherapy for prophylactic use or for controlled central nervous system (CNS) leukemia.
   2. Use of hydroxyurea for participants with rapidly proliferative disease is allowed before the start of study therapy and for the first 4 weeks on study treatment.
6. Recovery from non-hematologic toxic effects of prior treatment to Grade ≤1, or baseline value according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 classification (excluding infertility, alopecia, or Grade 1 neuropathy).
7. Baseline QT interval corrected using the Fridericia equation (QTcF) ≤ 480 msec. Note: This criterion does not apply to participants with a bundle branch block (BBB); for participants with BBB, a cardiology consult is recommended to ensure that QTcF is not prolonged.
8. Female participants who are women of childbearing potential (WOCBP) must have a negative serum or urine (beta-human chorionic gonadotropin (βhCG)) pregnancy test at screening and negative serum or urine test documented within the 24-hour period prior to the first dose of study drug. WOCBP are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression (Section 4.8.1).
9. Sexually active female participants who are WOCBP and male participants who are sexually active partners of WOCBP must agree to use a highly effective method of contraception during the course of the study from the date of informed consent and for at least 3 months after their last dose of study drug. Effective birth control methods include the following:

   1. Intrauterine device (IUD) plus one barrier method.
   2. Stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal).
   3. 2 barrier methods; effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).
   4. A vasectomized partner (where vasectomy was done at least 4 months prior to first dose of study treatment).
   5. True abstinence (ie, abstinence that is in line with the preferred and usual lifestyle of the participant).
10. Female and male participants must agree to refrain from egg/ova retrieval either for their own use or donation or from sperm donation, respectively, from the date of informed consent until 3 months after the last dose of study treatment.
11. Participant is willing and able to participate and comply with all study requirements and to provide signed and dated written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Relapsed/Refractory AML.
2. ELN (2022) favorable risk AML, except for nucleophosmin 1 (NPM1) mutated AML, which is allowed.
3. Acute promyelocytic leukemia (APL).
4. Positive Fms related receptor tyrosine kinase 3-Internal tandem duplication (FLT3-ITD) mutation.
5. Active CNS involvement by leukemia (other extramedullary disease is allowed).
6. Participants <18 years or >75 years of age.
7. Female participant who is pregnant or breastfeeding.
8. Participant plans to become pregnant or father a child (including ova or sperm donation) while enrolled in this study or within 3 months after last dose of study treatment (Section 4.8).
9. Participant has a known allergy or history of hypersensitivity to study drugs or their excipients.
10. Previous therapy with olutasidenib (or ivosidenib or other IDH1 inhibitor) or venetoclax (or another B cell lymphoma 2 (BCL-2) inhibitor).
11. Participant has active evidence of clinically significant unstable medical condition such as uncontrolled infection, severe metabolic abnormality, poorly controlled psychiatric illness, or symptomatic coronary artery disease (other than stable angina), which could place the participant at unacceptable risk of study treatment, per the Investigator's judgement.
12. Participants receiving treatment with strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors within 7 to 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Azoles are allowed with appropriate venetoclax dose reductions. Please note that participants receiving these medications would qualify for this study after undergoing a washout period of 7 to 14 days or 5 half-lives, whatever is longer for the inhibitor/inducer.
13. Participants receiving treatment with strong CYP3A inducers within 7 to 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Please note that participants receiving these medications would qualify for this study after undergoing a washout period of 7 to 14 days or 5 half-lives, whatever is longer for the inhibitor/inducer.
14. History of allogeneic hematopoietic stem cell transplant (HSCT) for a diagnosis other than AML if there is clinically significant active graft-versus-host disease (GVHD) or ongoing immunosuppressive therapy is required beyond prednisone 10 mg daily or equivalent. Otherwise, prior allogeneic HSCT is allowed.
15. Participants with a concurrent active malignancy under treatment.
16. Known history of active hepatitis B (HBV) or hepatitis C (HCV) infection or human immunodeficiency virus (HIV) infection (clinically detectable viral load).
17. Major surgery within 28 days prior to the first dose. Participants must have recovered from surgery and be without current complications.
18. Participants with impaired decision-making capacity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Excessive Toxicity | Up to 12 months
  The number of participants experiencing excessive toxicity in six (6) patient safety lead-in over the duration of study treatment will be reported. All treatment-emergent adverse events (TEAEs) will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Composite Complete Remission (CRc) | Up to 3 months
  Composite complete remission (CRc) among participants will be reported as a percentage. CRc is includes number of participants experiencing complete remission [CR], complete remission with partial hematologic recovery [CRh] or complete remission with incomplete hematologic recovery [CRi] after up to 3 cycles as defined by modified 2022 European LeukemiaNet (ELN) criteria.

SECONDARY OUTCOMES:
Number of Participants Experiencing Unacceptable Toxicity | Up to 13 months
  The number of participants experiencing unacceptable toxicity in entire cohort will be reported over the duration of study treatment. All toxicity will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of Participants Experiencing Treatment-Emergent Adverse Events | Up to 13 months
  The number of participants experiencing treatment-emergent adverse events (TEAEs) will be reported over the duration of study treatment. All toxicity will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of Participants Experiencing Serious Adverse Events | Up to 13 months
  The number of participants experiencing serious adverse events (SAEs) will be reported over the duration of study treatment. All toxicity will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of Participants Experiencing Adverse events of special interest (AESIs) | Up to 13 months
  The number of participants experiencing adverse events of special interest (AESIs) will be reported over the duration of study treatment. All toxicity will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of participants who died within 30-days | Up to 30 days
  The number of participants that die within 30-days after starting study therapy will be reported.
Number of participants who died within 60-days | Up to 60 days
  The number of participants that die within 60-days after starting study therapy will be reported.
Duration of Composite Complete Remission (CRc) | Up to 12 months
  Duration of CR over the duration of study treatment will be reported. Duration of CR is defined as time in months from CRc is first achieved until relapse, death, or off-study for other acute myeloid leukemia (AML) therapy.
Time to Composite Complete Remission (CRc) | Up to 12 months
  Time to composite complete remission (CRc) among participants will be reported in months. Time to CRc is defined is the period from Cycle 1 Day 1 (C1D1) to the date CRc is first achieved.
Percentage of Participants Receiving Allogeneic HCST | Up to 12 months
  The percentage of participants receiving allogenic stem cell transplant (HCST), over the duration of study treatment will be reported.
Percentage of Participants Achieving Complete Response (CR) | Up to 12 months
  The percentage of study participants achieving complete response (CR) to study treatment will be reported. Response will be assessed using on modified 2022 European LeukemiaNet (ELN) criteria for AML.
Overall Response Rate | Up to 12 months
  Overall response rate (ORR) (reported as a percentage), which includes complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete hematologic recovery (CRi), morphologic leukemia free state (MLFS), and partial response (PR) over the duration of study treatment, as defined by modified 2022 European LeukemiaNet (ELN) criteria.
Duration of response (DOR) | Up to 12 months
  Duration of response (DOR) over the duration of study treatment will be reported. The DOR is defined as the number of days from the date of initial response to the date of first documented disease progression/relapse or death, whichever occurs first.
Time to Response (TTR) | Up to 12 months
  Time to response (TTR) over the duration of study treatment will be reported in months. TTR is defined as the elapsed time from Cycle 1 Day 1 until complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete hematologic recovery (CRi), morphologic leukemia free state (MLFS), or partial response (PR) is first achieved.
Event-free survival (EFS) | Up to 12 months
  Event-free survival (EFS) among study participants over the duration of study treatment will be reported. EFS is defined as time in months from the date of treatment initiation (i.e., C1D1) to the date of documented treatment failure, relapse, or death from any cause, whichever occurs first, and will be calculated for all participants.
Overall survival (OS) | Up to 36 months
  Overall survival (OS) is defined as the elapsed time in months from the start of treatment until death from any cause. Alive participants will be censored at the last date known to be alive.
Minimal residual disease (MRD) negative rates | Up to 12 months
  Minimal residual disease (MRD) negative rates as assessed by multi-parameter flow cytometry (MPFC) and/or next generation sequencing (NGS)/polymerase chain reaction (PCR) based technology performed locally, will be reported as a percentage over the duration of study treatment.
Pharmacokinetics (PK): Cmax | Up to 9 months
  Maximum plasma concentration (Cmax) among study participants will be reported via the collection and analysis of blood samples. The peak concentration(Cmax) is the highest level of plasma concentration that occurs after drug administration.
Pharmacokinetics: Tmax | Up to 9 months
  Time to maximum plasma concentration (Tmax) among study participants will be reported via the collection and analysis of blood samples
Pharmacokinetics: Cmin | Up to 9 months
  Minimum plasma concentration (Cmin) among study participants will be reported via the collection and analysis of blood samples.
Pharmacokinetics: AUC | Up to 9 months
  Area under the plasma concentration-time curve (AUC)(0-24)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Watts, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No